CLINICAL TRIAL: NCT00691210
Title: Phase I Study of Vorinostat in Combination With Niacinamide, and Etoposide for the Treatment of Patients With Relapsed and Refractory Lymphoid Malignancies
Brief Title: Phase I Vorinostat in Combination With Niacinamide and Etoposide for Lymphoid Malignancies
Acronym: SAHA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAJ3001
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2015-03-10 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Hodgkin's Disease; Non-Hodgkin's Lymphoma
Keywords: Hodgkin's Disease; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Vorinostat; Niacinamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- V/N: Level 1 (Experimental): Vorinostat: 400mg Niacinamide: 20 mg/kg rounded to 100mg
  Interventions: Drug: Vorinostat; Drug: Niacinamide
- V/N: Level 2 (Experimental): Vorinostat: 400mg Niacinamide: 40 mg/kg rounded to 100mg
  Interventions: Drug: Vorinostat; Drug: Niacinamide
- V/N: Level 3 (Experimental): Vorinostat: 400mg Niacinamide: 60 mg/kg rounded to 100mg
  Interventions: Drug: Vorinostat; Drug: Niacinamide
- V/N: Level 4 (Experimental): Vorinostat: 400mg Niacinamide: 80 mg/kg rounded to 100mg
  Interventions: Drug: Vorinostat; Drug: Niacinamide
- V/N: Level 5 (Experimental): Vorinostat: 400mg Niacinamide: 100 mg/kg rounded to 100mg
  Interventions: Drug: Vorinostat; Drug: Niacinamide
- V/N/E: Level 1 (Experimental): Vorinostat: 400mg Niacinamide: 80 mg/kg rounded to 100mg Etoposide: 25 mg/m2
  Interventions: Drug: Vorinostat; Drug: Niacinamide; Drug: Etoposide
- V/N/E: Level 2 (Experimental): Vorinostat: 400mg Niacinamide: 80 mg/kg rounded to 100mg Etoposide: 50 mg/m2
  Interventions: Drug: Vorinostat; Drug: Niacinamide; Drug: Etoposide
- V/N/E: Level 3 (Experimental): Vorinostat: 400mg Niacinamide: 80 mg/kg rounded to 100mg Etoposide: 100 mg/m2
  Interventions: Drug: Vorinostat; Drug: Niacinamide; Drug: Etoposide

INTERVENTIONS:
Drug: Vorinostat — Dose escalation scheme (400 mg)
  Vorinostat is used to treat cutaneous T-cell lymphoma (CTCL, a type of cancer) in people whose disease has not improved, has gotten worse, or has come back after taking other medications. Vorinostat is in a class of medications called histone deacetylase (HDAC) inhibitors. It works by killing or stopping the growth of cancer cells.
  Other Names: SAHA
Drug: Niacinamide — Dose escalation scheme (20, 40, 60, 80, 100 mg/kg rounded to 100 mg)
  Niacinamide is a water soluble B-vitamin that has been evaluated for use in the treatment of pellagra, bullous pemphigoid, and as a radiation sensitizer in head and neck cancer.
  Other Names: Nicotinamide
Drug: Etoposide — Dose escalation scheme (0, 25, 50, 100 mg/m2)
  Etoposide is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug. This medication is classified as a "plant alkaloid" and "topoisomerase II inhibitor."
  Other Names: VP-16
  Arms: V/N/E: Level 1; V/N/E: Level 2; V/N/E: Level 3

SUMMARY:
The purpose of this study is to test the safety of a combination of two anticancer medicines, called vorinostat and etoposide, with a high dose of a vitamin called niacinamide. These medications will be tested at different dose levels. The investigators want to find out what effects, good and/or bad, it has on patients and their recurrent lymphoma. The first two drugs, vorinostat and niacinamide, suppress survival signals that lymphoma cells depend on. The third drug, etoposide can kill sensitive lymphoma cells alone or in combination with other chemotherapy drugs. Vorinostat is an anticancer agent that been approved by the Food and Drug Administration for use in cutaneous T-cell lymphoma. It is being evaluated in this study in combination with other anticancer medicines for use in other types of lymphoma. Vorinostat's use in combination with anticancer regimens is experimental. Niacinamide is a vitamin that is investigational or experimental when given at high doses as an anticancer agent. Niacinamide has not yet been approved by the Food and Drug Administration for use in lymphoma. Etoposide has been approved by the Food and Drug Administration for use in aggressive non-Hodgkin's lymphoma. However, the way it will be given in this clinical study is experimental.

DETAILED DESCRIPTION:
Subjects will be treated with vorinostat administered orally with daily dosing for 14 days of a 21-day treatment cycle in combination with niacinamide administered orally for 14 days in 21-day treatment cycle and etoposide administered intravenously on days 8,9 and 10 of a 21-day treatment cycle. Etoposide dose will be escalated until maximum tolerated dose (MTD) is determined.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed relapsed or refractory non-Hodgkin's lymphoma or Hodgkin's Disease (WHO criteria), for which they are unwilling or unable to undergo an autologous stem cell transplant
2. Must have received first line chemotherapy. No upper limit to number of prior therapies
3. Evaluable Disease
4. Age >18 years
5. Eastern Cooperative Oncology Group (ECOG) performance status <2
6. Life expectancy of greater than 3 months
7. Patients must have adequate organ and marrow function
8. Adequate Contraception
9. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Prior Therapy

   * Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
   * Patient is on any systemic steroids that have not been stabilized to the equivalent of ≤10 mg/day prednisone during the 7 days prior to the start of the study drugs
   * No monoclonal antibody within 3 months unless evidence of progression
2. Patients may not be receiving any other investigational agents
3. Patients with known central nervous system metastases, including lymphomatous meningitis
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat, niacinamide or etoposide
5. Uncontrolled intercurrent illness
6. Pregnant women
7. Nursing women
8. Active concurrent malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix). If there is a history of prior malignancy, the patient must be disease-free for ≥ 3 years
9. Patient is known to be Human Immunodeficiency Virus (HIV)-positive
10. Active Hepatitis A, Hepatitis B, or Hepatitis C infection
11. Patient has a history of surgery that would interfere with the administration or absorption of the oral study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2014-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Owen A O'Connor, MD, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Center for Lymphoid Malignancies at CUMC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amengual JE, Clark-Garvey S, Kalac M, Scotto L, Marchi E, Neylon E, Johannet P, Wei Y, Zain J, O'Connor OA. Sirtuin and pan-class I/II deacetylase (DAC) inhibition is synergistic in preclinical models and clinical studies of lymphoma. Blood. 2013 Sep 19;122(12):2104-13. doi: 10.1182/blood-2013-02-485441. Epub 2013 Aug 2. PMID 23913470

RESULTS

PARTICIPANT FLOW:
Groups:
- V/N: Level 2: Vorinostat: 400mg Niacinamide: 40 mg/kg rounded to 100mg
  Vorinostat (SAHA) and Niacinamide: dose escalation scheme
- V/N: Level 1: Vorinostat: 400mg Niacinamide: 20 mg/kg rounded to 100mg
  Vorinostat (SAHA) and Niacinamide: dose escalation scheme
- V/N: Level 3: Vorinostat: 400mg Niacinamide: 60 mg/kg rounded to 100mg
  Vorinostat (SAHA) and Niacinamide: dose escalation scheme
- V/N: Level 4: Vorinostat: 400mg Niacinamide: 80 mg/kg rounded to 100mg
  Vorinostat (SAHA) and Niacinamide: dose escalation scheme
- V/N: Level 5: Vorinostat: 400mg Niacinamide: 100 mg/kg rounded to 100mg
  Vorinostat (SAHA) and Niacinamide: dose escalation scheme
- V/N/E: Level 1: Vorinostat: 400mg Niacinamide: 80 mg/kg rounded to 100mg Etoposide: 25 mg/m2
  Vorinostat, Niacinamide and Etoposide: dose escalation scheme
- V/N/E: Level 2: Vorinostat: 400mg Niacinamide: 80 mg/kg rounded to 100mg Etoposide: 50 mg/m2
  Vorinostat, Niacinamide and Etoposide: dose escalation scheme
- V/N/E: Level 3: Vorinostat: 400mg Niacinamide: 80 mg/kg rounded to 100mg Etoposide: 100 mg/m2
  Vorinostat, Niacinamide and Etoposide: dose escalation scheme
Period: Overall Study
Arm/Group | V/N: Level 2 | V/N: Level 1 | V/N: Level 3 | V/N: Level 4 | V/N: Level 5 | V/N/E: Level 1 | V/N/E: Level 2 | V/N/E: Level 3
Started | 3 | 5 | 3 | 9 | 5 | 7 | 6 | 0
Completed | 3 | 5 | 3 | 6 | 5 | 6 | 6 | 0
Not Completed | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Not completed — Progression of Disease | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were no subjects enrolled or evaluable in VNE Level 3 Arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | V/N: Level 1 | V/N: Level 2 | V/N: Level 3 | V/N: Level 4 | V/N: Level 5 | V/N/E: Level 1 | V/N/E: Level 2 | V/N/E: Level 3 | Total
Number analyzed (Participants) | 5 | 3 | 3 | 9 | 5 | 7 | 6 | 0 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Between 18 and 65 years | 5 | 2 | 3 | 7 | 3 | 6 | 4 |  | 30
  >=65 years | 0 | 1 | 0 | 2 | 2 | 1 | 2 |  | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 4 | 2 | 2 | 2 |  | 15
  Male | 3 | 1 | 2 | 5 | 3 | 5 | 4 |  | 23

OUTCOME MEASURES:

1. Secondary Outcome: The Greatest Number of Cycles Received in Each Treatment Group
Description: The highest number of cycles received by an individual participant in the treatment groups. Each cycle was 21 days long.
Time Frame: up to 45 weeks
Measure: Number; unit: cycles
Groups:
- Vorinostat (SAHA) and Niacinamide: Level 1: Vorinostat: 400mg Niacinamide: 20 mg/kg rounded to 100mg
  Vorinostat (SAHA) and Niacinamide: dose escalation scheme
- Vorinostat (SAHA) and Niacinamide: Level 2: Vorinostat: 400mg Niacinamide: 40 mg/kg rounded to 100mg
  Vorinostat (SAHA) and Niacinamide: dose escalation scheme
- Vorinostat (SAHA) and Niacinamide: Level 3: Vorinostat: 400mg Niacinamide: 60 mg/kg rounded to 100mg
  Vorinostat (SAHA) and Niacinamide: dose escalation scheme
- Vorinostat (SAHA) and Niacinamide: Level 4: Vorinostat: 400mg Niacinamide: 80 mg/kg rounded to 100mg
  Vorinostat (SAHA) and Niacinamide: dose escalation scheme
- Vorinostat (SAHA) and Niacinamide: Level 5: Vorinostat: 400mg Niacinamide: 100 mg/kg rounded to 100mg
  Vorinostat (SAHA) and Niacinamide: dose escalation scheme
- Vorinostat, Niacinamide and Etoposide: Level 1: Vorinostat: 400mg Niacinamide: 80 mg/kg rounded to 100mg Etoposide: 25 mg/m2
  Vorinostat, Niacinamide and Etoposide: dose escalation scheme
- Vorinostat, Niacinamide and Etoposide: Level 2: Vorinostat: 400mg Niacinamide: 80 mg/kg rounded to 100mg Etoposide: 50 mg/m2
  Vorinostat, Niacinamide and Etoposide: dose escalation scheme
Arm/Group | Vorinostat (SAHA) and Niacinamide: Level 1 | Vorinostat (SAHA) and Niacinamide: Level 2 | Vorinostat (SAHA) and Niacinamide: Level 3 | Vorinostat (SAHA) and Niacinamide: Level 4 | Vorinostat (SAHA) and Niacinamide: Level 5 | Vorinostat, Niacinamide and Etoposide: Level 1 | Vorinostat, Niacinamide and Etoposide: Level 2
Number analyzed (Participants) | 5 | 3 | 3 | 6 | 5 | 6 | 5
cycles | 9 | 12 | 15 | 10 | 14 | 3 | 4

2. Secondary Outcome: The Number of Dose Delays and Reductions at the MTD
Time Frame: continuous
Reporting Status: Not Posted

3. Secondary Outcome: The Prevalence of Anti-tumor Activity
Time Frame: continuous
Reporting Status: Not Posted

4. Secondary Outcome: Pharmacodynamic Markers of Target Effect in Paired Tissue Biopsies
Time Frame: continuous
Reporting Status: Not Posted

5. Primary Outcome: The Maximum Tolerated Dose (MTD) of Niacinamide in the Combination of Vorinostat and Niacinamide
Time Frame: 3 years
Population: There were no evaluable patients at these levels.
Measure: Number; unit: mg/kg
Groups:
- Vorinostat (SAHA) and Niacinamide: Level 1-5: Vorinostat: 400mg Niacinamide: 20-100 mg/kg rounded to 100mg
  Vorinostat (SAHA) and Niacinamide: dose escalation scheme
- Vorinostat, Niacinamide and Etoposide: Level 1-2: Vorinostat: 400mg Niacinamide: 80 mg/kg rounded to 100mg Etoposide: 25-50 mg/m2
  Vorinostat, Niacinamide and Etoposide: dose escalation scheme
Arm/Group | Vorinostat (SAHA) and Niacinamide: Level 1-5 | Vorinostat, Niacinamide and Etoposide: Level 1-2
Number analyzed (Participants) | 22 | 0
mg/kg | 100 |

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 30 days post end of treatment for each patient
Description: Adverse events were collected by patient reporting and physical exam with an attending and graded using Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0).
Arm/Group | Vorinostat (SAHA) and Niacinamide: Level 1 | Vorinostat (SAHA) and Niacinamide: Level 2 | Vorinostat (SAHA) and Niacinamide: Level 3 | Vorinostat (SAHA) and Niacinamide: Level 4 | Vorinostat (SAHA) and Niacinamide: Level 5 | Vorinostat, Niacinamide and Etoposide: Level 1 | Vorinostat, Niacinamide and Etoposide: Level 2
Serious Adverse Events (participants affected / at risk) | 2/5 | 1/3 | 0/3 | 5/9 | 3/5 | 2/7 | 1/6
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 3/3 | 9/9 | 5/5 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (SAHA) and Niacinamide: Level 1 (N=5) | Vorinostat (SAHA) and Niacinamide: Level 2 (N=3) | Vorinostat (SAHA) and Niacinamide: Level 3 (N=3) | Vorinostat (SAHA) and Niacinamide: Level 4 (N=9) | Vorinostat (SAHA) and Niacinamide: Level 5 (N=5) | Vorinostat, Niacinamide and Etoposide: Level 1 (N=7) | Vorinostat, Niacinamide and Etoposide: Level 2 (N=6)
Acidosis (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALT (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
AST (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver Failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Uric Acid (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nausea (General disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DVT (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand-Foot Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leg Weakness & Numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Soreness in mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MSSA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chord Compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphotemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Low CO2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urea Nitrogen (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (SAHA) and Niacinamide: Level 1 (N=5) | Vorinostat (SAHA) and Niacinamide: Level 2 (N=3) | Vorinostat (SAHA) and Niacinamide: Level 3 (N=3) | Vorinostat (SAHA) and Niacinamide: Level 4 (N=9) | Vorinostat (SAHA) and Niacinamide: Level 5 (N=5) | Vorinostat, Niacinamide and Etoposide: Level 1 (N=7) | Vorinostat, Niacinamide and Etoposide: Level 2 (N=6)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 5 (11) | 2 (8) | 1 (2) | 0 (0)
2 episodes of feeling weak & unbalanced (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
3 Puncatate skin Leasions on Arm(mosquito bites) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Abdominal Cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acid Reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (following RT) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitated/Irritable Mood (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alk Phos (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALT (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 1 (2) | 2 (4) | 1 (1) | 1 (2) | 0 (0)
Ammonia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANC (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (7) | 2 (3) | 2 (9) | 0 (0)
Anesthesia of Forehead (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (4) | 2 (3) | 7 (14) | 2 (2) | 3 (5) | 3 (4)
Anxiety (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Armpit Burning (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspergillus fumigatus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AST (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 1 (2) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Bacterial SuperInfections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bad Taste in Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Belching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilateral Lower Extremity Edema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood in Stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bloodshot eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body Aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning near rectum (likely zoster related) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bumps on Tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation in throat (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burning with Urination (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calf Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (lesion on knee) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central Disc Herniation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Chest Pressure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHF Exacerbation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 1 (1) | 0 (0)
Clear Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clots in Urine (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Collapsed Lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 2 (4) | 3 (4) | 4 (7) | 2 (3) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 2 (5) | 4 (10) | 4 (9) | 2 (2) | 0 (0)
Cramping (intermittent) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cramping (menopausal symptoms) (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cramping in Hands & Feet (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Blood and lymphatic system disorders) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
D-Dimer (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decrease in Strength (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decrease in taste (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decrease Sex Drive (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 2 (7) | 7 (12) | 3 (6) | 1 (3) | 1 (3)
Difficulty initiating urinary stream (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diffuse Erythematous Rash ( extremeties) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diffuse PapilarRash ( hypersensitivity reaction) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Discomfort in Stomach (pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disseminated Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dry Eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Heaving (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Lips (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
DVT ( Left subclavala vein) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (DOE) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 4 (6) | 2 (4) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear Ache (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 2 (2) | 0 (0)
Elevated Base Excess (intermittent) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated Creatinine (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (7) | 1 (1) | 0 (0)
Elevated Lactate (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Elevated pH (intermittent) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated PO2 (intermittent) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated WBC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (mild & intermittent) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythematous (slightly on neck) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eschai of ight index finger (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial Tingling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (Metabolism and nutrition disorders) | 1 (1) | 2 (7) | 3 (9) | 9 (17) | 5 (17) | 4 (9) | 2 (2)
Fever (Metabolism and nutrition disorders) | 1 (3) | 2 (5) | 2 (4) | 4 (6) | 4 (4) | 2 (2) | 1 (1)
Finger Parasthesias (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 2 (5) | 3 (3) | 0 (0)
Gagging (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gas (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
General Malaise (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GERD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin Swelling (post -op site) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gums/Teeth tender feeling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand- Foot Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headaches (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 5 (11) | 2 (9) | 1 (2) | 0 (0)
Heart Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoptysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hoarse Voice (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperactive (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperactivity of the Gut (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphatemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Hypothermia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Infections and infestations (Bacterium gram neg rods) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INR (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
itching (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Joint Aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lack of Concentration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leakage from rectum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left Breast Itchy Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left Eye Redness (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left Groin Lymph Node Pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Left lower quadrant abdominal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left Nipple Bump (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left Sided Abdominal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left Upper Quandrant Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leg Weakness/numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Legs Cramps (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Light Headedness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Liver Dysfunction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver Failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low Chloride (intermittent) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Low CO2 (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Low PCO2 (intermittent) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Low PO2 (intermittent) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower Neck Tighness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MAPS (in 50's) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic Acidosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metallic Taste (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Mild Dyspena (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mild Hypovalemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mild Increase in Tremor (in off week) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mild Increasein Intention Tremor (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mild Neck Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mild Right Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mild Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth Sore (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular Pain(Buttocks to toes) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (12) | 3 (5) | 8 (28) | 5 (21) | 5 (10) | 3 (5)
Neck Aches (site of enlarged LN) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (8) | 2 (3) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Neutropenic Spesis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Night Sweats (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 1 (1) | 0 (0)
Nosebleed (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
O2 saturation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocassional Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Occasional sweating at night (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Occational lightheadedness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odor with Urination (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Papular Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Parasthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Petechiae Hard Palate (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Probable) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Port Infections and infestations (staphylococcus species, coagulase negative) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post Nasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncopal Episode (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritic Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (4) | 0 (0) | 1 (1)
Ptosis of the right eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulled Back Muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (mid area of chest) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash(below left breast) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash(blotchy dry spots on hands) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Redness & slight bump on right of nose (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Hip Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Arm Swelling(bug bite) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Cheek Red Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Eye Redness (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Foot Cramp (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right Hand Inflammation(cat scratch) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Leg Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Lower Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right Lower Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right rib Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right Shoulder Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right Side Mouth Sore (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Upper Quadrant Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rigors (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal and Penile Edema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensory Neuropathy in feet (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 1 (3) | 1 (1) | 0 (0)
Short-term memory loss (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Headache (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Lesion lower back (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin tenderness on face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Slight cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Slight dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Slight Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Slight hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore Foot(stepped on nail) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore Lymph Nodes(w/ pain) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (5) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Soreness in mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soreness of gumlike (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphyloccus aureus (MSSA) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stiff Fingers (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach Cramps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach Virus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Strong Odor of Urine (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suprapubic pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sweating (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swollen Cheeks (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swollen Glands (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swollen Hands & Feets (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
T6/7 & T9/10 Cord Compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (3) | 0 (0)
Taste Changes (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
T-Cell Lymphoproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenderness in Mouth, Esophagus, Stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat Tightening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (6) | 2 (3) | 1 (2) | 2 (4) | 1 (1) | 1 (4) | 0 (0)
Toe Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toe Parasthesias (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trace Edema (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Transient Viral Infections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulcerations in mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respitatory Infections and infestations (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Upper/Mild Back Spams (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upset Stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urea Nitrogen (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Urgency with urination (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URI (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uric Acid (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTI (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaginal dryness (menopausal symptoms) (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomitiing (Gastrointestinal disorders) | 1 (1) | 2 (10) | 2 (3) | 6 (24) | 4 (7) | 2 (3) | 1 (1)
Weak urine stream (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wide based gait when walking (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Yeast Infections and infestations (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Zoster (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (5) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes